CLINICAL TRIAL: NCT01040468
Title: Lifestyle Intervention Versus Bariatric Surgery for Type 2 Diabetes
Brief Title: Surgery Or Lifestyle Intervention for Type 2 Diabetes (SOLID)
Acronym: SOLID
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 809984; 1RC1DK086132 (NIH)
Record Dates: First submitted 2009-12-24; First posted 2009-12-29 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Bariatric Surgery; Roux-en-Y Gastric Bypass; Gastric Banding; Obesity; Weight loss; Insulin sensitivity; GLP-1; Meal Challenge; Euglycemic Clamp
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity; Weight Loss; Insulin Resistance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Roux-en-Y Gastric Bypass surgery (Active Comparator): Surgical intervention for weight loss
  Interventions: Procedure: Roux-en-Y Gastric Bypass surgery
- Laparoscopic Adjustable Gastric Banding surgery (Active Comparator): Surgical intervention for weight loss
  Interventions: Procedure: Laparoscopic Adjustable Gastric Banding surgery
- Intensive Lifestyle Modification (Active Comparator): Lifestyle intervention for weight loss
  Interventions: Behavioral: Intensive Lifestyle Modification

INTERVENTIONS:
Procedure: Roux-en-Y Gastric Bypass surgery — Surgical intervention for weight loss. This is a one-year study and participants will attend five study visits.
  Arms: Roux-en-Y Gastric Bypass surgery
Procedure: Laparoscopic Adjustable Gastric Banding surgery — Surgical intervention for weight loss. This is a one-year study and participants will attend five study visits.
  Arms: Laparoscopic Adjustable Gastric Banding surgery
Behavioral: Intensive Lifestyle Modification — Intensive lifestyle modification program for weight loss. Participants randomized to this condition will receive an weekly individual treatment of 30 minutes for the first 6 months and every-other-week sessions from months 7 to 12. Treatment will be provided by a behavioral psychologist or registered dietitian following a structured curriculum used in our prior studies. During the first 4 months, participants will be prescribed a 1000-1200 kcal/d diet that provides four daily servings of meal replacement products (liquid shakes, cereals, meal bars, etc), combined with an evening dinner entree. Each serving of the meal replacement (HMR 170; Boston, MA) will provide 170 calories, with 16 g of protein, 22 g of carbohydrate, and 2 g of fat. Dinner entrees (containing at least 20 g of protein and approximately 220-260 kcal) will be consumed with a garden salad and a serving of fruit (and other vegetables allowed ad libitum throughout the day).
  Arms: Intensive Lifestyle Modification

SUMMARY:
This research study will investigate the safety and effectiveness of weight loss surgery for overweight persons with type 2 diabetes. Eligible patients will undergo one of 2 types of weight loss surgery, Roux-en-Y gastric bypass, or laparoscopic adjustable gastric banding, or an intensive lifestyle modification. Participants will be closely followed for one year to compare the effects of these treatments on diabetes remission.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 65 years old.
* Diagnosis of type 2 diabetes.
* Individuals with a BMI of 30-40 kg/m2
* Approval for bariatric surgery (as confirmed by medical evaluation)
* Insurance coverage for bariatric surgery
* Willingness to change diet, physical activity and weight.
* Ability to communicate with the investigator and be legally competent, provide written informed consent.

Exclusion Criteria:

* Diagnosis of type 1 diabetes, diagnosis of maturity-onset diabetes of the young (MODY), or latent autoimmune diabetes in adults (LADA) (all of which are associated with ß-cell destruction), daily insulin requirements > 100 units, and poor preoperative glycemic control, as indicated by a HbA1c > 6.5 - ≤ 8.5 or HbA1c > 8.6 - < 9.5 (individuals with this HbA1c value will require medical clearance and approval from the study physician).
* Children and adolescents are not eligible to participate in the study.
* Pregnant women (or those who intend to become pregnant during the study period) and women who are currently breastfeeding are not eligible to participate.
* Use of medications known to significantly increase body weight, such as chronic systemic steroids or certain psychiatric medications (e.g., lithium tricyclic antidepressants and anti-psychotic agents).
* Non-ambulatory individuals, defined as those who are unable to walk at least one city block without a cane or walker.
* Any major illnesses that the surgical team believes present too great a risk for surgery. These include severe cardiac and pulmonary diseases, as well as uncontrolled type 2 diabetes.
* Evidence of major depression or other psychiatric disorder (schizophrenia, bipolar disorder, major depression, bulimia nervosa, etc.) that is uncontrolled, poorly controlled, or, in the opinion of the Investigators, significantly interferes with daily living and functioning.
* Any current (past 12 months) substance abuse or dependence disorder.
* Participants with moderate anemia (Hgb < 12 mg/dl for men and Hgb < 11 mg/dl for women)
* Conditions that may falsely elevate or decrease HbA1c values, including hemolytic or iron-deficiency anemia, hemoglobinopathies, and uremia.
* Abnormal laboratory tests which are clinically significant per the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2009-09; Primary Completion 2015-03 (Actual); Study Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
The primary objective of this study is to compare the rates of diabetes remission over one year. | One year

SECONDARY OUTCOMES:
Secondary objectives of this study are to determine the effects of the three treatment conditions on insulin sensitivity, endogenous glucose production, postprandial insulin release, and levels of gut hormones (including GLP-1). | One year
To compare other benefits (e.g., improvements in quality of life, dietary intake, and physical activity), as well as risks (e.g., hypoglycemia, cholecystitis, early and late surgical complications), of the three interventions. | One year
To examine the attitudes that patients, health care professionals, and insurance providers have toward the use of bariatric surgery to treat type 2 diabetes. | One year

CONTACTS AND LOCATIONS:
Overall Officials: David B Sarwer, Ph.D., Principal Investigator — University of Pennsylvania; Thomas A Wadden, Ph.D., Principal Investigator — University of Pennsylvania; Noel Williams, M.D., Principal Investigator — University of Pennsylvania Department of Surgery
Locations (1):
- University of Pennsylvania Center for Weight and Eating Disorders, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Center for Weight and Eating Disorders website — http://www.med.upenn.edu/weight/research.shtml
- See also: Bariatric Surgery Program at Penn website — http://www.pennmedicine.org/bariatrics/